CLINICAL TRIAL: NCT00070239
Title: A Phase I Clinical, Pharmacokinetic and Pharmacodynamic Study of Flavopiridol in Patients With Refractory Solid Tumors and Hematologic Malignancies
Brief Title: Alvocidib in Treating Patients With Metastatic or Unresectable Refractory Solid Tumors or Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00039; NCI-2009-00039 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 03-082; P 6052; CDR0000331689; 03-082 (Other: Dana-Farber Cancer Institute); 6052 (Other: CTEP); U01CA062490 (NIH)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Hematopoietic/Lymphoid Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Hematologic Neoplasms | interventions — alvocidib; Fluorodeoxyglucose F18; alovudine; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

ARMS (1):
- Treatment (Experimental): PART 1 (closed to accrual as of 8/2005): Patients receive alvocidib IV over 1 hour on days 1, 8, and 15.
  Cohorts of 3-6 patients receive escalating doses of alvocidib until the MTD* is determined.
  PART 2: Patients receive alvocidib IV over 1 hour at or below the MTD determined in part 1 and then receive a maintenance dose of alvocidib IV over 1-6 hours on days 1, 8, and 15. Cohorts of 3-6 patients receive escalating durations of the maintenance dose of alvocidib until the MTD* is determined. An additional cohort of 10-20 patients receives alvocidib over 1 hour on days 1 and 15 at the MTD.
  NOTE: *The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  In both parts, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alvocidib; Other: pharmacological study; Radiation: fludeoxyglucose F 18; Other: fluorine F 18 fluorothymidine; Procedure: positron emission tomography

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Radiation: fludeoxyglucose F 18 — Correlative studies
  Other Names: 18FDG; FDG
Other: fluorine F 18 fluorothymidine — Correlative studies
  Other Names: 18F-FLT; 3'-deoxy-3'-[18F]fluorothymidine; fluorothymidine F-18
Procedure: positron emission tomography — Correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed

SUMMARY:
This phase I trial is studying the side effects and best dose of alvocidib in treating patients with metastatic or unresectable refractory solid tumors or hematologic malignancies. Drugs used in chemotherapy, such as alvocidib, work in different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the maximum tolerated dose of flavopiridol in patients with metastatic or unresectable refractory solid tumors or hematologic malignancies. (Accrual for patients with hematologic malignancies temporarily closed as of 11/30/04)

SECONDARY OBJECTIVES:

I. Determine the safety profile and toxic effects of this drug in these patients.

II. Determine the pharmacokinetics of this drug in these patients. III. Determine, by pharmacodynamic assays, the ability of this drug to inhibit cyclin-dependent kinase activity in tumor tissue, normal proliferating tissues, circulating tumor cells, and in plasma in these patients.

IV. Determine, preliminarily, the antitumor activity of this drug in these patients.

OUTLINE: This is a 2-part, dose-escalation, multicenter study.

PART 1 (closed to accrual as of 8/2005): Patients receive alvocidib IV over 1 hour on days 1, 8, and 15.

Cohorts of 3-6 patients receive escalating doses of alvocidib until the maximum tolerated dose (MTD)* is determined.

PART 2: Patients receive alvocidib IV over 1 hour at or below the MTD determined in part 1 and then receive a maintenance dose of alvocidib IV over 1-6 hours on days 1, 8, and 15. Cohorts of 3-6 patients receive escalating durations of the maintenance dose of alvocidib until the MTD* is determined. An additional cohort of 10-20 patients receives alvocidib over 1 hour on days 1 and 15 at the MTD.

NOTE: *The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

In both parts, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 month and then every 2 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy, including the following types:

  * Hematologic malignancy, including any of the following: (Accrual for patients with hematologic malignancies temporarily closed as of 11/30/04)
  * Mantle cell lymphoma
  * Morphologically confirmed disease
  * CD20 and CD5 positive
  * Any other refractory lymphoma
  * Chronic lymphocytic leukemia
* Rai stage III or IV and meeting at least 1 of the following criteria for active disease:

  * Weight loss > 10% in the last 6 months
  * Fatigue
  * Fever or night sweats with no evidence of infection
  * Progressive anemia or thrombocytopenia
  * Progressive lymphocytosis with a lymphocyte doubling time of < 6 months
  * Marked hypogammaglobulinemia or paraproteinemia
  * Progressive splenomegaly and/or lymphadenopathy
  * Multiple myeloma
  * Disease confirmed by bone marrow aspirate and/or biopsy
  * Relapsed or refractory disease after the most recent treatment regimen
  * Quantifiable monoclonal immunoglobulin in serum and/or urine
* Solid tumor, including but not limited to any of the following:

  * Breast cancer
  * Histologically or cytologically confirmed stage IV invasive disease
  * HER-2 positivity not required for study enrollment
  * Tumor overexpressing HER-2 should be confirmed by immunohistochemistry OR fluorescence in situ hybridization
  * Small cell lung cancer
  * Extensive stage or limited stage disease in relapse
  * Extrapulmonary small cell carcinoma allowed
  * Squamous cell carcinoma of the head and neck
  * Metastatic, recurrent, or refractory disease
  * Renal cell carcinoma
  * Mesothelioma
  * Pleural or peritoneal disease of epithelial, sarcomatoid, or mixed subtype
  * Melanoma
  * Kaposi's sarcoma
  * Metastatic or unresectable disease for which standard therapy does not exist or is no longer effective
  * Measurable or nonmeasurable disease (solid tumor patients)
  * Measurable disease defined as at least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or 10 mm by spiral CT scan
* Nonmeasurable disease includes any of the following:

  * All other lesions, including lesions < 20 mm by conventional techniques or 10 mm by spiral CT scan
  * Bone lesions
  * Cytologically positive pleural or peritoneal disease
  * Elevated tumor marker (e.g., CEA, CA 125, CA 19-9, or other tumor marker)
  * Multinodular or confluent nonmeasurable pulmonary, hepatic, adrenal, intra-abdominal, or skin metastases
  * Previously treated with at least 1 chemotherapy regimen*
  * Prior therapy may have included combined modality treatment (e.g., full-dose chemotherapy and radiotherapy with radiosensitizing chemotherapy)
  * Prior therapy with flavopiridol allowed provided the patient was enrolled in a flavopiridol clinical trial employing a different schedule NOTE: *Except in cases where chemotherapy is not known to be effective (e.g., renal cell carcinoma, chondrosarcoma, or gastrointestinal stromal tumor)
  * No active CNS metastases
* History of CNS metastases allowed provided all of the following criteria are met:

  * Previously treated and stable and asymptomatic for at least 4 weeks since the completion of treatment
  * Image documentation required
  * Off steroids or on a stable dose of steroids for at least 1 week
* Hormone receptor status:

  * Not specified
* Age

  * 18 and over
* Sex

  * Male or female
* Menopausal status

  * Not specified
* Performance status

  * ECOG 0-1 OR
  * Karnofsky 70-100%
* Life expectancy

  * More than 12 weeks
* Hematopoietic

  * Absolute neutrophil count > 1,000/mm^3*
  * Platelet count > 75,000/mm^3 (50,000 for hematologic malignancies)* (Accrual for patients with hematologic malignancies temporarily closed as of 11/30/04) NOTE: *Unless abnormality is caused by tumor burden and not cumulative prior chemotherapy
* Hepatic

  * Bilirubin normal
  * AST/ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Renal

  * Creatinine ≤ 2.0 mg/dL OR
  * Creatinine clearance ≥ 60 mL/min
* Cardiovascular

  * No myocardial infarction within the past 6 months
  * No unstable angina within the past 6 months
  * No transient ischemic attack or cerebrovascular accident within the past 6 months
  * No history of arterial vascular events
  * No new cardiac arrhythmias likely to be related to cardiac ischemia within the past 6 months
  * No symptomatic congestive heart failure
* Pulmonary

  * No history of pulmonary embolism within the past 6 months
* Gastrointestinal

  * No chronic diarrheal disease within the past 6 months
  * No severe malnutrition
  * No intractable emesis
* Other

  * Not pregnant or nursing
  * Negative pregnancy test
  * Fertile patients must use effective hormonal or barrier contraception
  * No ongoing or active infection
  * No other concurrent uncontrolled illness
  * No psychiatric illness or social situation that would preclude study compliance
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* At least 3 weeks since prior radiotherapy No prior radiotherapy to 50% or more of bone marrow
* Recovered from all prior therapy No other concurrent investigational agents No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-08; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days
MTD (or recommended phase II dose), defined as one dose level below that which produces two instances of DLT during the first 28-day course and the level at which no more than one of six patients experiences DLT during course 1 | 28 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters, including maximum concentration (Cmax), half-life, area under the curve (AUC), clearance, and volume of distribution | 24 hours, 48 hours, 72 hours, and 8 weeks
  Determined by nonlinear regression analysis of geometric mean plasma profile. Cmax in patients w/stable disease or response at 8 weeks compared to those who progressed using Mann-Whitney test. Wilcoxon signed-rank test to compare concentration and metabolic ratios directly following infusion and 24, 48, 72 hrs later. Concentration and metabolic ratios compared in patients w/ and w/o toxicities of diarrhea, neutropenia, and asthenia using Mann- Whitney test. Fisher's exact test to assess association of flavopiridol systemic metabolism (low vs. high metabolic ratio) w/development of toxicity.
Potency of alvocidib in plasma based on change in proliferation of stimulated peripheral blood mononuclear cells (PBMCs) | Baseline to up to 72 hours of day 1 course 1
Change in tumor metabolism and proliferation assessed by fludeoxyglucose F 18 (FDG) and fluorine F 18 fluorothymidine (FLT) positron emission tomography (PET) | Baseline to up to day 19 of course 2
  Each type of pre- and post-treatment scans may be analyzed as paired data. The FDG and FLT data will be correlated to explore the relationship between tumor metabolism and tumor proliferation, for example, using Pearson or Spearman correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Shapiro, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States